CLINICAL TRIAL: NCT03965221
Title: Comparison of Men's Prevention Apps to Research Efficacy
Acronym: COMPARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Public Health Foundation Enterprises, Inc. (Other)
Collaborators: Adolescent Trials Network for HIV/AIDS Interventions (Network); Adolescent and Young Adult Research (AYAR), CORE Center (Unknown); Children's Hospital of Philadelphia (Other); Baylor College of Medicine (Other); University of South Florida (Other); Emory University (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Fenway Community Health (Other); San Francisco Department of Public Health (Other Government); University of North Carolina, Chapel Hill (Other); The Children's Hospital at Montefiore (CHAM) (Unknown); National Institute on Drug Abuse (NIDA) (NIH); National Institute of Mental Health (NIMH) (NIH); Brown University (Other); RAIN, Inc. (Unknown)
Responsible Party: Principal Investigator, Albert Liu, Director, Clinical Research, Public Health Foundation Enterprises, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 19-0260; 5U19HD089881 (NIH)
Record Dates: First submitted 2019-05-17; First posted 2019-05-28 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: HIV/AIDS; Sexually Transmitted Diseases; Pre-exposure Prophylaxis; Risk Reduction
Keywords: PrEP; HIV Testing; Sexually Transmitted Infections; Mobile app; Young men who have sex with men; Technology
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Sexually Transmitted Diseases; Risk Reduction Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- LYNX (Experimental): LYNX is developed using IMB model and engages youth through entering sexual diary data, earning badges, and calculating a personalized sexual protection (Sex Pro) score, which informs and motivates youth around HIV/STI testing and PrEP uptake. Behavioral skills are built through HIV/STI testing reminders, presenting options for home HIV testing and/or linkage to nearby testing services, and access to an online chat with support for HIV/STI testing and PrEP referral.
  Interventions: Behavioral: LYNX
- MyChoices (Experimental): MyChoices is adapted from an app for adult MSM, HealthMindr, developed using SCT. The app aims to increase HIV testing and PrEP uptake by increasing self- regulation, self-reflection, and self-efficacy around HIV testing and PrEP uptake. Brief surveys about sexual risk and protective health behaviors within the app are used to assist users in tracking and self-monitoring their behaviors and creating a personalized HIV testing plan. Quizzes, videos and infographics as well as "Help me Choose," "Ordering," and geofencing functions are used to maximize self-efficacy around HIV prevention and uptake of PrEP.
  Interventions: Behavioral: MyChoices
- Standard of Care (No Intervention): Provision of referrals to local HIV/STI testing and PrEP resources.

INTERVENTIONS:
Behavioral: LYNX — Access to the LYNX mobile app which includes the Sex Pro score tool, sex diary, badges, PrEP information and video testimonials, HIV/STI testing reminders and geo-location features, and asynchronous chat feature.
  Arms: LYNX
Behavioral: MyChoices — Access to the MyChoices mobile app which includes the HIV test plan with reminders, STI information, PrEP resources, links to testing and PrEP sites, and geo-location features.
  Arms: MyChoices

SUMMARY:
A randomized three arm control trial to examine the efficacy of two distinct apps (LYNX and MyChoices) developed for young men who have sex with men (YMSM) compared to standard of care (SOC) information about HIV testing and PrEP (Pre-Exposure Prophylaxis).

DETAILED DESCRIPTION:
COMPARE is part of the iTech NIH U19, which has an overall goal to develop innovative technology-focused interventions addressing the HIV prevention and care continuum for youth. In years 1-2 of the iTech grant, the investigators optimized and pilot tested using a similar study design and identical study outcomes, two distinct mobile apps called LYNX and MyChoices. Each app is designed to increase HIV testing and PrEP uptake among YMSM. In this study, the individual apps are being tested in this follow-on research study to evaluate for efficacy. YMSM will be randomized to receive either MyChoices, LYNX, or SOC. LYNX uses the Information-Motivation-Behavior Skills (IMB) model and is a highly interactive mobile app to promote accurate risk perception, increase HIV/STI testing, and linkage to PrEP. MyChoices is guided by the Social Cognitive Theory (SCT) model, is adapted from HealthMindr and developed using iterative feedback from youth refined to maximize acceptability among YMSM. It includes three major functions that are designed to promote self-efficacy, self-regulation, goal-setting and environmental influences to impact behavior change. The SOC includes information on HIV testing and PrEP with the provision of referrals to local HIV/STI testing and PrEP resources.

ELIGIBILITY:
Inclusion Criteria:

* 15 to 29 years.
* Assigned male sex at birth and male identified.
* Self-report being HIV uninfected or HIV status-unknown at screening.
* Self-report having not had an HIV test in the past 3 months.
* Self-report not currently taking PrEP.
* Self-report at least one episode of anal intercourse with a male or transfemale partner during the last 12 months.
* Able to understand, read, and speak English.
* Owns or leases a phone with Android platform or iOS platform, has an active data plan Has phone setting in English or Spanish, or willing to use an English or Spanish phone setting over the course of the study (Spanish setting is only for bilingual participants who speak both English and Spanish fluently)
* Willing and able to attend an in-person baseline study visit in one of the study site areas, or willing to attend a remote online baseline study visit

Exclusion Criteria:

* Currently enrolled in another HIV intervention study.
* Prior enrollment in an HIV vaccine trial with receipt of experimental vaccine product.
* Enrollment in Aims 2 and 3 of the prior MyChoices (UNC IRB# 17-0256) or LYNX (UNC IRB# 17-0170) studies
* Any medical, psychiatric, or social condition or other responsibilities that, in the judgment of the investigator, would make participation in the study unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives.
* Not willing and/or not able to download the MyChoices and LYNX apps onto their phone

Ages: 15 Years to 29 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Cisgender men
Enrollment: 381 (Actual)
Dates: Start 2019-10-14 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Efficacy for HIV testing: Proportion who complete >= 1 HIV test | 6 months post baseline
  Proportion who complete >= 1 HIV test
Efficacy for PrEP uptake: Proportion who uptake PrEP | 6 months post baseline
  Proportion who uptake PrEP
Efficacy for STI testing: Proportion who complete >=1 STI test | 6 months post baseline
  Proportion who complete >=1 STI test

SECONDARY OUTCOMES:
Efficacy for HIV testing: Proportion who complete >= 1 HIV test | 12 months post baseline
  Proportion who complete >= 1 HIV test
Efficacy for PrEP uptake: Proportion who uptake PrEP | 12 months post baseline
  Proportion who uptake PrEP
Efficacy for STI testing: Proportion who complete >=1 STI test | 12 months post baseline
  Proportion who complete >=1 STI test

CONTACTS AND LOCATIONS:
Overall Officials: Albert Y Liu, MD, MPH, Principal Investigator — San Francisco Department of Public Health; Katie B Biello, PhD, MPH, Principal Investigator — Brown University
Locations (8):
- United States (8):
  - University of South Florida, Infectious Diseases, Tampa, Florida
  - PRISM Health, Atlanta, Georgia
  - Ayar @ Core, Chicago, Illinois
  - Fenway Health Center, Boston, Massachusetts
  - Montefiore Children's Hospital, The Bronx, New York
  - RAIN, Inc, Charlotte, North Carolina
  - Adolescent Initiative at Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Baylor College of Medicine, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
Raw data will be available to outside individuals through contacting the multiple principal investigators (MPIs) at two different times. The first will be after all of the baseline data is collected. The investigators will institute a concept plan process where internal study staff first have the availability to write primary papers or give presentations on particular topics. After this, if outside individuals wish to analyze data, the investigators will welcome this collaboration. A similar process will happen for outcome data; however this will not be possible until the publication and release of the outcome paper(s). Information regarding the availability of data for analysis will be listed on the MPIs' web pages. Contact information for the MPIs will be listed in all manuscripts and publications as another means to access data.

REFERENCES:
- [Derived] Biello KB, Mayer KH, Scott H, Valente PK, Hill-Rorie J, Buchbinder S, Ackah-Toffey L, Sullivan PS, Hightow-Weidman L, Liu AY. The Effects of MyChoices and LYNX Mobile Apps on HIV Testing and Pre-Exposure Prophylaxis Use by Young US Sexual Minority Men: Results From a National Randomized Controlled Trial. JMIR Public Health Surveill. 2025 Feb 5;11:e63428. doi: 10.2196/63428. PMID 39908084